CLINICAL TRIAL: NCT00766961
Title: Randomized Comparison of Trans-catheter Arterial Embolization (TAE) and Surgery in Patients With Major Peptic Ulcer Bleeding Uncontrolled by Endoscopic Therapy
Brief Title: TAE and Surgery in Patients With Peptic Ulcer Bleeding Uncontrolled by Endoscopic Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Karolinska University Hospital (Other); Erasme University Hospital (Other); King Chulalongkorn Memorial Hospital (Other)
Responsible Party: Principal Investigator, James Yun-wong Lau, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TAE
Record Dates: First submitted 2008-10-03; First posted 2008-10-06 (Estimated); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: Peptic Ulcer; Bleeding
Keywords: Peptic ulcer bleeding uncontrolled by endoscopic therapy.
MeSH Terms: conditions — Peptic Ulcer; Hemorrhage | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TAE group (Active Comparator): Trans-catheter arterial embolization
  Interventions: Procedure: Trans-catheter arterial embolization
- Surgery group (Active Comparator): Surgery
  Interventions: Procedure: Surgery

INTERVENTIONS:
Procedure: Trans-catheter arterial embolization — Trans-catheter arterial embolization
  Other Names: TAE
  Arms: TAE group
Procedure: Surgery — Surgery
  Arms: Surgery group

SUMMARY:
The aim of the study is to compare the outcomes of trans-catheter arterial embolization (TAE) and surgery as salvage therapy of peptic ulcer bleeding after failed endoscopic therapy.

DETAILED DESCRIPTION:
The aim of the study is to examine the hypothesis that trans-catheter arterial embolization (TAE) is safer than and probably as effective as surgery in the control of bleeding from ulcers after failed endoscopic therapy. Patients with major arterial bleeding that cannot be stopped by endoscopic therapy will be randomly assigned to receive immediate TAE or surgery. Primary outcome will be death within 30 days of randomization. Secondary outcomes include recurrent bleeding after assigned treatment, need for additional intervention either in the form of interventional radiology or surgery, and post procedural morbidities.

ELIGIBILITY:
Inclusion Criteria:

* Patients with bleeding peptic ulcers documented during endoscopic therapy AND anyone of the following:
* Forrest I bleeding that fails to be controlled by therapy during first endoscopy
* Check endoscopy after clinical re-bleeding of Forrest I bleeding
* Forrest IIa or an initial IIb but a sizable artery unveiled upon clot elevation in a high risk ulcer defined by:
* posterior bulbar duodenal ulcer > 2cm, or
* an angular notch / lesser curve gastric ulcer > 5cm that fail an attempt at endoscopic therapy together with evidence of a significant bleed (hypotension with SBP < 90mmHg, fresh hematemesis or hematochezia).

Exclusion Criteria:

* Refusal to participate in trial
* No consent
* Age < 18
* Pregnancy
* Moribund patients
* Patients with terminal malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2007-04; Primary Completion 2017-03 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Mortality within 30 days of randomization | 30 days
  Mortality within 30 days of randomization

SECONDARY OUTCOMES:
Recurrent bleeding after assigned treatment | 60 days
  Recurrent bleeding after assigned treatment
The need for additional intervention either in the form of interventional radiology | 60 days
  The need for additional intervention either in the form of interventional radiology
Post procedural morbidities | 60 days
  Post procedural morbidities
The need for additional intervention either in the form of surgery | 60 days
  The need for additional intervention either in the form of surgery

CONTACTS AND LOCATIONS:
Overall Officials: James YW LAU, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Endoscopy Center, Prince of Wales Hospital, Hong Kong, China